CLINICAL TRIAL: NCT03640962
Title: Investigation of the Relationship in Sleep With Low Back Pain in Postmenopausal Period
Brief Title: Relationship in Sleep With Low Back Pain in Postmenopausal Period
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Other Study IDs: IBU17.02.2015/28-210
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Postmenopausal Symptoms
Keywords: Postmenopause; Low back pain; Woman
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation — This cross-sectional study was conducted in 368 postmenopausal women aged between 40 and 65 years. This study was carried out in family health centers in Istanbul. Data were collected via face-to-face interviews by the researchers.

SUMMARY:
Introduction:The aim of this study was to investigate the incidence of low back pain in postmenopausal period and the relationship between low back pain and emotional state,sleep and quality of life i aimed at investigating low back pain during postmenopausal period of women and its correlation with the emotional state,sleep quality and the quality of life of woman.

Method:This cross-sectional study was conducted in 368 postmenopausal women aged between 40 and 65 years.All participants were recorded frequency and severity of low back pain,depressive symptoms and anxiety,quality of life and sleep quality.Outcome measures are described in more detail below.

DETAILED DESCRIPTION:
Participants This cross-sectional study was conducted in 368 postmenopausal women aged between 40 and 65 years. This study was carried out in family health centers in Istanbul. Participants who have not had menstrual bleeding for the last 1 year and, with FSH levels above 30 mlU / ml were included in this study. My exclusion criteria in the study were illiterate women. All participants were given informed consent about the aim and methods of the study.

Study design Data were collected via face-to-face interviews by the researcher. Socio-demographic data ascertained included age, Body Mass Index (BMI), marital status, tobacco and alcohol use, medication use, presence of chronic disease, age of menopause onset, and educational level. All participants were recorded frequency and severity of low back pain, depressive symptoms, anxiety, quality of life and sleep quality. Outcome measures are described in more detail below. According to the power analysis results, when the number of enough participants was reached, the study was stopped. Ethics committee approval for the study was obtained from the Istanbul Science University Ethics Committee for Clinical Researches (IBU17.02.2015/28-210).

Outcome measurements Pain To determine the frequency of current pain, all eligible participants were evaluated and asked to report whether they had had pain. All participants were evaluated for severity of pain using an 11-point numeric visual analog scale (VAS; 0= no pain; 10=worst pain imaginable). Participants were asked to characterize their pain severity along a horizontal, 10-cm line. Participants were questioned about the severity of low back pain during rest, during activity and at night. Statistics were made by categorizing the severity of low back pain during rest, activityand at night. Low back pain intensity were classified that according to the cut-off point of the VAS. (0.1-3.8 mild pain, 3.9-5.7 moderate pain, 5.8-10 severe pain).

Emotional Status Hospital Anxiety and Depression Scale (HADS) was used to determine the level of anxiety and depression of the participants. It contains 14 items, seven related to depression and seven to anxiety. Each item is rated in a 4 point scale. A subscale score of 0-21 and to a total score of 0-42. Scores of 11 or more on either sub-scale is considered to be a significant "case" of psychological morbidity, while scores of 8 to 10 represent "borderline" and 0 to 7 "normal". It was originally developed in 1983 by Zigmond and Snaith in order to evaluate the risk for anxiety and depression in patient and to measure the level and severity of anxiety/ depression. The validity and reliability of Turkish version of the HAD Scale was tested in 1997 by Aydemir.

Quality of Life Nottingham Health Profile (NHP) was used to determine quality of life of the participants. NHP is a general health status scale (health-related quality of life), which aims to measure a patient's perceived emotional, social and physical health status. This scale consists of 38 items formed as yes-no questions that cover 6 subscales of the quality of life. These six subscales are sleep (5 item), energy level (3 item), emotional status (9 item), social isolation (5 item), physical mobility (8 item) and pain (8 item). Each section is scored from 0-100. 0 indicates the best health status, 100 indicates the worst health status. In the study, the sub-scores of NHP and total NHP scores were evaluated. Total NHP score was obtained from the sum of the sub-scores. The scale was developed by Hunt et al.(1981). NHP is an easy-to-use scale and the validity and reliability of Turkish version was by Küçükdeveci at al.(2000).

Sleep Quality Pittsburgh Sleep Quality Index (PSQI) was used to determine sleep quality of the participants. PSQI was originally developed by Buysse et al.(1989). PSQI was adapted into Turkish by Ağargün et al.(1996). PSQI is consisting of 24 items, 19 of which are self-assessment questions and the rest 5 are answered by patient's spouse or roommate. The scored 18 items covers 7 components, namely subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping medication and daytime dysfunction. Each component is evaluated on a 0-3 interval scale whereby 3 reflect the negative extreme on the Likert Scale. The total score obtained from the seven components are equivalent to the total scale score. The total score ranges between 0 and 21; higher scores indicate worse sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have not had menstrual bleeding for the last 1 year
* FSH levels above 30 mlU / ml

Exclusion Criteria:

* illiterate women

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Study Population: Postmenopausal women aged between 40 and 65 years. This study was carried out in family health centers in Istanbul.
Sampling Method: Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-09-22 (Estimated)

PRIMARY OUTCOMES:
Pain of low back pain: Visual Analog Scale | 1 minute
  Visual Analog Scale: To determine the frequency of current pain, all eligible participants were evaluated and asked to report whether they had had pain. All participants were evaluated for severity of pain using an 11-point numeric visual analog scale (VAS; 0= no pain; 10=worst pain imaginable). Participants were asked to characterize their pain severity along a horizontal, 10-cm line. Participants were questioned about the severity of low back pain during rest, during activity and at night. Statistics were made by categorizing the severity of low back pain during rest, activityand at night. Low back pain intensity were classified that according to the cut-off point of the VAS. (0.1-3.8 mild pain, 3.9-5.7 moderate pain, 5.8-10 severe pain)

SECONDARY OUTCOMES:
Emotional status: Hospital Anxiety and Depression Scale | 5 minutes
  Hospital Anxiety and Depression Scale (HADS) was used to determine the level of anxiety and depression of the participants. It contains 14 items, seven related to depression and seven to anxiety. Each item is rated in a 4 point scale. A subscale score of 0-21 and to a total score of 0-42. Scores of 11 or more on either sub-scale is considered to be a significant "case" of psychological morbidity, while scores of 8 to 10 represent "borderline" and 0 to 7 "normal". It was originally developed in 1983 by Zigmond and Snaith in order to evaluate the risk for anxiety and depression in patient and to measure the level and severity of anxiety/ depression. The validity and reliability of Turkish version of the HAD Scale was tested in 1997 by Aydemir
Quality of life of women: Nottingham Health Profile | 5 minutes
  Nottingham Health Profile (NHP) was used to determine quality of life of the participants. NHP is a general health status scale (health-related quality of life), which aims to measure a patient's perceived emotional, social and physical health status. This scale consists of 38 items formed as yes-no questions that cover 6 subscales of the quality of life. These six subscales are sleep (5 item), energy level (3 item), emotional status (9 item), social isolation (5 item), physical mobility (8 item) and pain (8 item). Each section is scored from 0-100. 0 indicates the best health status, 100 indicates the worst health status. In the study, the sub-scores of NHP and total NHP scores were evaluated. Total NHP score was obtained from the sum of the sub-scores. The scale was developed by Hunt et al.(1981). NHP is an easy-to-use scale and the validity and reliability of Turkish version was by Küçükdeveci at al.(2000)
Sleep quality: Pittsburgh Sleep Quality Index | 5 minutes
  Pittsburgh Sleep Quality Index (PSQI) was used to determine sleep quality of the participants. PSQI was originally developed by Buysse et al.(1989). PSQI was adapted into Turkish by Ağargün et al.(1996). PSQI is consisting of 24 items, 19 of which are self-assessment questions and the rest 5 are answered by patient's spouse or roommate. The scored 18 items covers 7 components, namely subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping medication and daytime dysfunction. Each component is evaluated on a 0-3 interval scale whereby 3 reflect the negative extreme on the Likert Scale. The total score obtained from the seven components are equivalent to the total scale score. The total score ranges between 0 and 21; higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: TOMRIS DUYMAZ, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomris Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided